CLINICAL TRIAL: NCT05204160
Title: Phase II Study of Pembrolizumab as Salvage Therapy Among Multiple Myeloma Patients Progressing on CAR-T Cell Therapy
Brief Title: Pembrolizumab as Salvage Therapy for the Treatment of Multiple Myeloma in Patients Progressing on CAR-T Cell Therapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Emory University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ajay Nooka, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003182; NCI-2021-08718 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship5388-21 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2022-01-11; First posted 2022-01-24 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (pembrolizumab) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies the effect of pembrolizumab in treating patients with multiple myeloma that is growing, spreading, or getting worse (progressing) on chimeric antigen receptor (CAR)-T cell therapy. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of pembrolizumab in patients who have received B- cell maturation antigen (BCMA)-directed adoptive cell therapy (ACT) and have clinical evidence of progression.

II. To obtain anti-tumor activity (best response rates: objective response rate [ORR], very good partial response, [VGPR], complete response [CR], stringent complete remission [sCR], minimal response disease [MRD] negativity) in patients treated with pembrolizumab.

SECONDARY OBJECTIVES:

I. To evaluate the expansion of engrafted T cells following pembrolizumab administration in the peripheral blood and within the tumor microenvironment.

II. To evaluate the phenotype and function of engrafted T cells following pembrolizumab administration.

III. Progression free survival (PFS) and overall survival (OS) among patients progressing after ACT that received pembrolizumab.

IV. To determine immunogenicity of the salvage regimen.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject is, in the investigator's opinion, willing and able to comply with the protocol requirements
* Subject has given voluntary signed written informed consent before performance of any study-related procedure that is not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to their future medical care
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1
* Have documented multiple myeloma as defined by the International Myeloma Working Group (IMWG) 2014 criteria including: Clonal bone marrow plasma cells >= 10% (If bone marrow has less than 10% clonal plasma cells, more than one bone lesion is required to distinguish from solitary plasmacytoma with minimal marrow involvement). In addition, the patient must meet one of the criteria in c1 or c2:

  * Evidence of end organ damage that can be attributed to the underlying plasma cell proliferative disorder, specifically (one or more of the following):

    * Hypercalcemia: serum calcium > 0.25 mmol/L (> 1 mg/dL) higher than the upper limit of normal (ULN) or > 2.75 mmol/L (> 11 mg/dL)
    * Renal insufficiency: Creatinine clearance (CrCl) < 40 mL/min (measured or estimated by validated equations) or serum creatinine > 177 umol/L (> 2 mg/dL)
    * Anemia: hemoglobin value of > 20 g/L below the lower limit of normal, or a hemoglobin value < 100 g/L
    * Bone lesions: 1 or more osteolytic lesions on skeletal radiography, computed tomography (CT), or magnetic resonance imaging (MRI) (Clonality should be established by showing kappa/lambda-light-chain restriction on flow cytometry, immunohistochemistry, or immunofluorescence. Bone marrow plasma cell percentage should preferably be estimated from a core biopsy specimen; in case of a disparity between the aspirate and core biopsy, the highest value should be used)
  * Any one or more of the following:

    * Clonal bone marrow plasma cell percentage >= 60% (Clonality should be established by showing kappa/lambda-light-chain restriction on flow cytometry, immunohistochemistry, or immunofluorescence. Bone marrow plasma cell percentage should preferably be estimated from a core biopsy specimen; in case of a disparity between the aspirate and core biopsy, the highest value should be used)
    * Involved: uninvolved serum free light chain (FLC) ratio > 100 (These values are based on the serum Freelite assay. The involved FLC must be >= 100 mg/L
    * > 1 focal lesions on MRI studies; Each focal lesion must be 5 mm or more in size
* Measurable disease as defined by any of the following:

  * Serum M-protein level >= 1.0 g/dL or urine M-protein level >= 200 mg/24 hours
  * IgA, IgD, IgE, or IgM multiple myeloma: serum M-protein level >= 0.5 g/dL or urine M-protein level >= 200 mg/24 hours; or
  * Light chain multiple myeloma without measurable disease in the urine: serum Ig free light chain (FLC) >= 10 mg/dL and abnormal serum Ig kappa/lambda FLC ratio
* Must have undergone BCMA-directed CART cell therapy and have evidence of progression per IMWG criteria upon response assessment
* Must have at least 4-week washout period for all the investigational monoclonal antibodies
* Men and women, age >= 18 years or legal age of consent per local regulations (whichever is greater)
* Female patients who:

  * Are postmenopausal for at least 1 year before the screening visit, OR
  * Are surgically sterile, OR
  * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
  * Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting study drugs
* Male patients, even if surgically sterilized (ie, status post-vasectomy), must agree to one of the following:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 4 weeks after the last dose of study drug, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)

Exclusion Criteria:

* Renal insufficiency, defined as creatinine clearance =< 30 mL/min (either actual or calculated value), within 21 days of initiation of protocol therapy. The Cockcroft - Gault formula should be used for calculating creatinine clearance values
* Platelet count =< 75,000 cells/mm^3 at time of screening evaluation. Platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days before study enrollment
* Participants with an absolute neutrophil count (ANC) =< 1000 cells/mm^3 at time of screening evaluation. Growth factors may not be used to meet ANC eligibility criteria within 14 days of obtaining screening evaluation
* Participants with hemoglobin level < 7.5 g/dL, at time of screening. Transfusion may not be used to meet eligibility criteria within 7 days of obtaining screening evaluation
* Participant had undergone ACT > 12 weeks from study enrollment
* Participants with hepatic impairment, defined as bilirubin >= 1.5 x institutional upper limit of normal (ULN) or aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]), alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]), or alkaline phosphatase >= 3x institutional ULN
* Patients may be receiving concomitant therapy with bisphosphonates and low dose corticosteroids (e.g., prednisone up to but no more than 10 mg orally [p.o.] once daily [q.d.] or its equivalent) for other rheumatological manifestations. Doses of corticosteroid should be stable for at least 7 days prior to study treatment.)
* Known significant cardiac abnormalities including:

  * Congestive heart failure, New York Heart Association (NYHA) class III or IV
  * Uncontrolled angina, arrhythmia or hypertension
  * Myocardial infarction within the past six months
  * Any other uncontrolled or severe cardiovascular condition
* Prior cerebrovascular event with residual neurologic deficit
* Serious, intercurrent illness including, but not limited to, clinically relevant active infection, known active hepatitis B or C viral infection, known human immunodeficiency virus (HIV) infection, uncontrolled diabetes mellitus, or serious co-morbid medical conditions such as chronic restrictive pulmonary disease, and cirrhosis
* Any condition, including laboratory abnormalities, that in the opinion of the investigator places the subject at unacceptable risk if he/she were to participate in the study
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection
* Known hypersensitivity to acyclovir or similar anti-viral drug
* Participants with known central nervous system (CNS) involvement
* Female participants pregnant or breast-feeding
* Participants who have undergone major surgery =< 4 weeks prior to starting study drug or who have not recovered from side effects of the surgery
* Participants with any significant history of non-compliance to medical regimens or unwilling or unable to comply with the instructions given to him/her by the study staff
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol
* Participation in other clinical trials, including those with other investigational agents not included in this trial, within 30 days of the start of this trial and throughout the duration of this trial
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Has severe hypersensitivity to (grade >= 3) to pembrolizumab and/or any of its excipients
* Subjects that have undergone prior allogeneic stem cell transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-02-27 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 3 years
  The ORR is defined as the proportion of treated subjects who achieve a best response of minimal residual disease negativity, complete response (CR), stringent (s)CR, very good partial response, or partial response using the International Myeloma Working Group criteria. The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Proportion of patients achieving stable disease or better will also be reported at 6 months and 12 months; Response rates will be reported along with 95% confidence intervals will be estimated using the Clopper-Pearson method. Chi-square test will be used to compare the efficacy in term of tumor response rate between the different groups.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 3 years
  For progression free survival, progression or death from any cause will be defined as the event. PFS rate of two patient groups stratified by dose levels or response status will be estimated with the Kaplan-Meier method and compared using the log-rank test, respectively. Cox proportional hazards models will be further used in the multivariable analyses to assess adjusted effect of dose levels on the patients' PFS after adjusting for other factors
Overall survival (OS) | Up to 3 years
  For overall survival, death from any cause will be defined as the event. OS rate of two patient groups stratified by dose levels or response status will be estimated with the Kaplan-Meier method and compared using the log-rank test, respectively. Cox proportional hazards models will be further used in the multivariable analyses to assess adjusted effect of dose levels on the patients' OS after adjusting for other factors
Immunogenicity of the salvage regimen | Up to 3 years
  Will evaluate the efficacy of the salvage regimen from a clinical and immunological aspect to determine the benefit it provides among patients who have received BCMA-directed adoptive cell therapy (ACT) and have clinical evidence of progression. Depending on whether data is normally distributed, t-test or Wilcoxon rank sum test will be used to compare each biomarker between any two groups stratified by dosage, response, or other factors, respectively. General linear model (GLM) will be used to compare each biomarker between multiple dose levels with and without adjusting for other factors. Logistics regression model will be further employed to test the adjusted effect of biomarker on the response rate after adjusting for dosage as well as other factors.
Incidence of adverse events (AEs) | Up to 3 years
  Proportion of acute (at 3 weeks, evaluation prior to next cycle) and late toxicity (beyond 6 months) will be reported, and 95% confidence intervals will be estimated using the Clopper-Pearson method. Adverse events will be graded using Common Terminology Criteria for Adverse Events (version 4.03). Any occurrence and severe (worst grade >= 3) AEs will be tabulated.

CONTACTS AND LOCATIONS:
Overall Officials: Ajay K Nooka, MD,MPH,FACP, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States